CLINICAL TRIAL: NCT00460382
Title: Prospective Clinical Trial to Assess Safety and Efficacy of DRV/r(TMC 114/r), ETV(TMC 125) and MK-0518 in Addition to OBT in HIV-1 Infected Patients With Limited to No Treatment Options ANRS 139 TRIO
Brief Title: Clinical Trial to Assess the Efficacy of Darunavir/Ritonavir (DRV/r), Etravirine (ETV) and Raltegravir (MK-0518) in HIV Patients With Resistant Viruses
Acronym: ANRS139 TRIO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry); Janssen-Cilag Tibotec (Unknown)
Responsible Party: French National Agency for Research on AIDS and Viral Hepatitis, French National Agency for Research on AIDS and Viral Hepatitis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-000670-23; ANRS 139 TRIO
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: HIV Infections
Keywords: HIV infections; HIV integrase inhibitor; etravirine; darunavir; MK 0518; raltegravir; Treatment Experienced; Antiviral drug resistance
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Darunavir; Ritonavir; etravirine; Enfuvirtide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: raltegravir potassium — 400 mg twice a day
  Other Names: Isentress
Drug: darunavir/ritonavir — 2 pills of 300 mg twice a day
  Other Names: Prezista
Drug: etravirine — 2 pills of 100 mg twice a day
  Other Names: TMC125
Drug: Optimized background regimen — NRTIs and or enfuvirtide (investigator choice)
  Other Names: OBT; enfuvirtide

SUMMARY:
The purpose of this study is to look at the safety and efficacy of a combination of 3 new antiretroviral drugs: darunavir, etravirine and MK-0518 (raltegravir) in patients who have multi-resistant viruses and limited treatment options. An optimized background regimen that may include nucleoside reverse transcriptase inhibitors (NRTIs) and enfuvirtide can be added, if possible, to this combination. Patients will undergo treatment for 48 weeks and virological efficacy will be evaluated at week 24.

DETAILED DESCRIPTION:
Methods: A phase II pilot, prospective, open label, single arm multicentric clinical trial assessing a darunavir/ritonavir, etravirine and MK-0518-containing regimen, if possible associated to an optimized background regimen that may include NRTIs and enfuvirtide, in HIV-1 infected patients failing combination antiretroviral therapy with multi-resistant viruses.

Treatment strategy: Patients will receive raltegravir (MK-0518), darunavir/ritonavir (TMC114/r) and etravirine (TMC125) and if possible an optimized background therapy.

* raltegravir (MK-0518) (400 mg x 2/d = one 400 mg pill twice daily)
* darunavir (600 mg x 2/d= two 300 mg pills twice daily with meal)
* ritonavir (100 mg x 2/d = one 100 mg pill twice daily with meal)
* etravirine (200 mg x 2/d = two 100 mg pills twice daily with meal)
* if possible an optimized background therapy: may include NRTI(s) and enfuvirtide but not nonnucleoside reverse transcriptase inhibitors (NNRTIs) and protease inhibitors (PIs). NRTIs choice is left to the clinician's discretion. Enfuvirtide is highly recommended in enfuvirtide-naive patients but is left to the clinician.

Main outcome: proportion of patients with HIV RNA levels of less than 50 copies/ml in an intent to treat analysis at W24.

Secondary outcomes: proportions of patients with HIV RNA levels of less than 50 copies/ml at week 48, with HIV RNA levels of less than 400 copies/ml at week 24 and 48; HIV RNA level evolution between baseline and week 48; HIV proviral DNA and 2LTR circle HIV DNA between baseline and week 48; number and type of resistance mutations in case of virologic failure occurrence; CD4 lymphocyte count and proportion evolution between baseline and week 48; HIV infection progression; frequency of the study regimen modifications and interruption; study regimen tolerance; study regimen adherence; association between study drugs' minimum concentrations at week 4 and virologic success at week 24; evolution of pharmacokinetic parameters of study drugs between week 1 and week 4 in the Pharmacokinetic substudy.

Sample size: 103 patients

Enrollment period: 24 weeks

Patient's participation duration: 52 weeks

An extended follow-up (from week 52 to week 96) has been added in April 2008.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and above
* Documented HIV-1 infection.
* History of virological failure on NNRTIs (patients with a history of toxicity to nevirapine and efavirenz may be enrolled in this study).
* On a combination antiretroviral therapy for at least 8 weeks prior to the screening visit (if on tipranavir, or enfuvirtide these drugs should have been introduced more than 8 weeks before the screening visit).
* Patient naive to darunavir, etravirine and to integrase inhibitors
* Plasma viral load at screening visit over 1000 copies/ml, (no CD4 restriction).
* Genotypic resistance testing at the screening visit:

  * Protease inhibitor mutations: over or equal to 3 primary protease inhibitor mutations among: D30N, V32I, L33F, M46I/L, I47A/V, G48V, I50L/V, I54M, L76V, V82A/F/L/T/S, I84V, N88S and L90M (IAS list 2006) but below or equal to 3 mutations among the following: V11I, V32I, L33F, I47V, I50V, I54L/M, G73S, L76V, I84V et L89V (virus sensitivity to darunavir/ritonavir).
  * Reverse transcriptase mutations: over or equal to 3 NRTI mutations (among IAS list) and below or equal to 3 mutations among: A98G, L100I, K101Q/P/E, K103H/N/S/T, V106A/M, V108I, E138G/K/Q, V179D/E/F/G/I, Y181C/I/V/C/H/L, Y188C/H/L, G190A/C/E/Q/S, P225H, F227C/L, M230I/L, P236L, K238N/T and Y318F (virus sensitivity to etravirine)

Exclusion Criteria:

* Non effective barrier contraception in women of child bearing potential
* Pregnant women or women who are breastfeeding
* Opportunistic infection at the acute phase
* Decompensated cirrhosis (stage B or C of Child-Pugh score)
* Malignancy requiring chemotherapy or radiotherapy
* Contraindicated medications being taken by the patient (listed in protocol)
* Allergy to the active substances and expedients of darunavir, etravirine and raltegravir.
* Haemoglobin < 7g/dl, neutrophil cell count < 500/mm3, platelets < 50,000/mm3, creatinine clearance < 50 ml/mn, P. alkaline, AST, ALT or total bilirubin over or equal to 3 times normal values.
* Patients receiving experimental agents with an exclusion period for participation in other studies applicable at the screening visit of the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HIV RNA levels of less than 50 copies/ml in an intent to treat analysis at week 24 | week 24

SECONDARY OUTCOMES:
Proportions of patients with HIV RNA levels of less than 50 copies/ml at week 48, with HIV RNA levels of less than 400 copies/ml at weeks 24 and 48 | week 24 and 48
HIV RNA level evolution between baseline and week 48 | from week 0 to 48
HIV proviral DNA and 2LTR circle HIV DNA between baseline and week 48 | from week 0 to 48
Number and type of resistance mutations in case of virologic failure occurrence | from week 0 to 48
CD4 lymphocyte count and proportion evolution between baseline and week 48 | from week 0 to 48
HIV infection progression | from week 0 to 48
Frequency of the study regimen modifications and interruption | from week 0 to 48
Study regimen tolerance | from week 0 to 48
Study regimen adherence | from week 0 to 48
Association between study drugs' minimum concentrations at week 4 and week 12 and virologic success at week 24 | from week 4 to 24
Evolution of pharmacokinetics parameters of study drugs in the PK substudy | betwwen week 1 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Yazdan YAZDANPANAH, MD PHD, Principal Investigator — Hôpital Tourcoing FRANCE; Geneviève CHENE, MD PHD, Study Director — INSERM U897 BORDEAUX FRANCE
Locations (1):
- Hôpital Gustave Dron, Service Maladies Infectieuses, Tourcoing, France